CLINICAL TRIAL: NCT02147054
Title: Pilot Study - Assessing the Impact of Using a Neuromuscular Blocking Agent to Reduce Neuromuscular Junction Damage and Intermediate Syndrome in Organophosphorus (OP) Insecticide Poisoned Patients Requiring Ventilation
Brief Title: A Pilot Study Using Rocuronium to Prevent Intermediate Syndrome After Organophosphorus Insecticide Poisoning
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Peradeniya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rocuronium Pilot May 14
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-10

CONDITIONS: Organophosphate Poisoning
Keywords: Organophosphate poisoning; Intermediate syndrome; Rocuronium
MeSH Terms: conditions — Organophosphate Poisoning | interventions — Rocuronium; Sugammadex

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rocuronium with >95% inhibition (Active Comparator): IV Rocuronium to be given:
  * Bolus dose of Rocuronium 0.3 mg/kg to achieve >95% inhibition as indicated by Train of Four monitoring
  * Continuous infusion of 1.5 mg/kg/hr to maintain level of inhibition
  * To continue until two rises in butyrylcholinesterase seen or for a maximum of 5 days
  Interventions: Drug: Rocuronium; Drug: Sugammadex
- Rocuronium with 50% inhibition (Active Comparator): IV Rocuronium to be given:
  * Bolus dose of Rocuronium 0.3 mg/kg to achieve 50% inhibition as indicated by Train of Four monitoring
  * Continuous infusion of 1.5 mg/kg/hr to maintain level of inhibition
  * To continue until two rises in butyrylcholinesterase seen or for a maximum of 5 days
  Interventions: Drug: Rocuronium; Drug: Sugammadex
- No Rocuronium (No Intervention): No Rocuronium will be given

INTERVENTIONS:
Drug: Rocuronium
  Other Names: Esmeron
  Arms: Rocuronium with 50% inhibition; Rocuronium with >95% inhibition
Drug: Sugammadex — Effect of Rocuronium will be reversed at the appropriate time using Sugammadex 16mg/kg as a single dose which may be repeated once.
  Other Names: Bridion
  Arms: Rocuronium with 50% inhibition; Rocuronium with >95% inhibition

SUMMARY:
Organophosphate pesticide poisoning causes close to 300 000 deaths per year worldwide. Many patients who ingest organophosphates require ventilation; of these patients approximately 50% die. Much of the mortality in these ventilated patients is secondary to intermediate syndrome. This is because OP pesticides inhibit acetylcholinesterase, causing an excess of acetylcholine at nerve synapses and the neuromuscular junction (NMJ). At the NMJ, the excess acetylcholine causes overstimulation and damage, which may lead to sudden respiratory arrest or prolonged ventilation and its associated complications.

The investigators believe that blocking these receptors using a neuromuscular blocking agent such as Rocuronium will protect the NMJ from damage and thus prevent intermediate syndrome and reduce number of intubated days and mortality.

In this pilot randomised controlled trial Rocuronium, a competitive nicotinic receptor antagonist, will be used to bind to the receptor at the neuromuscular junction and to block the effects of the accumulated acetylcholine. The effects of OP pesticide on cholinesterase in the blood will then be monitored and Rocuronium withdrawn using Sugammadex as the OP is eliminated from the body.

DETAILED DESCRIPTION:
Primary outcome: Number of days intubated

ELIGIBILITY:
Inclusion criteria:

* Male or female
* Age over 16
* Clinical diagnosis of OP insecticide poisoning
* Admission to Intensive Care Unit for Ventilation
* Informed consent from family
* Train of four measurement > 50%

Exclusion criteria:

* Age 16 or under
* Pregnant
* Consent not obtained from patient or patient's family

Ages: 17 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of intubated days | Upto 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Indika Gawarammana, MD FRCPE PhD, Principal Investigator — South Asian Clinical Toxicology Research Collaboration; Michael Eddleston, MA PhD FRCP, Study Director — University of Edinburgh; Vasanti Pinto, MD FRCA FCARSCI, Study Director — University of Peradeniya; Vajira Weerasinghe, BDS MPhil PhD, Study Director — University of Peradeniya
Locations (1):
- Peradeniya Teaching Hospital, Peradeniya, Central Province, Sri Lanka

IPD SHARING:
Plan to Share IPD: No